CLINICAL TRIAL: NCT04570033
Title: The Utility of 18F-fluorocholine PET/CT in the Imaging of Parathyroid Adenomas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Military Institute od Medicine National Research Institute (Other)
Collaborators: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Andrzej Mazurek, MD PhD, Military Institute od Medicine National Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Military Institute of Medicine
Record Dates: First submitted 2020-09-21; First posted 2020-09-30 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Hyperparathyroidism; Parathyroid Adenoma
Keywords: PET/CT; fluorocholine
MeSH Terms: conditions — Hyperparathyroidism; Parathyroid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- patients with hyperparathyroidism (Experimental): We prospectively enrolled 65 consecutive patients with primary hyperparathyroidism (PHPT) who underwent neck ultrasound (US) and parathyroid scintigraphy (99mTc/99mTc-MIBI dual phase). Twenty-two patients had unsuccessful parathyroid surgery prior to the study
  Interventions: Diagnostic Test: We assessed sensitivity of 18F-FCH PET/CT in preoperative localisation of hyperfunctioning parathyroid tissue in patients with primary hyperparathyroidism

INTERVENTIONS:
Diagnostic Test: We assessed sensitivity of 18F-FCH PET/CT in preoperative localisation of hyperfunctioning parathyroid tissue in patients with primary hyperparathyroidism — We prospectively enrolled 65 consecutive patients with PHPT who underwent neck ultrasound (US) and parathyroid scintigraphy (99mTc/99mTc-MIBI dual phase). Twenty-two patients had unsuccessful parathyroid surgery prior to the study. PET/CT scans were performed 65.0 ± 13.3 min after injection of 218.5 ± 31.9 MBq of 18F-fluorocholine (FCH). Three experienced nuclear medicine physicians assessed the detection rate of hyperfunctioning parathyroid tissue. Response to parathyroidectomy and clinical follow-up served as a reference test. Per-patient sensitivity and positive predictive value (PPV) were calculated for patients who underwent surgery.

SUMMARY:
We assessed sensitivity of 18F-FCH PET/CT in preoperative localisation of hyperfunctioning parathyroid tissue in patients with primary hyperparathyroidism (PHPT).

DETAILED DESCRIPTION:
We prospectively enrolled 65 consecutive patients with PHPT who underwent neck ultrasound (US) and parathyroid scintigraphy (99mTc/99mTc-MIBI dual phase). Twenty-two patients had unsuccessful parathyroid surgery prior to the study. PET/CT scans were performed 65.0 ± 13.3 min after injection of 218.5 ± 31.9 MBq of 18F-fluorocholine (FCH). Three experienced nuclear medicine physicians assessed the detection rate of hyperfunctioning parathyroid tissue. Response to parathyroidectomy and clinical follow-up served as a reference test. Per-patient sensitivity and positive predictive value (PPV) were calculated for patients who underwent surgery.

ELIGIBILITY:
Inclusion Criteria:

* primary hyperparathyroidism and neck US and the dual-phase 99mTc/99mTc-MIBI SPECT/CT scintigraphy performed prior to the PET/CT scan

Exclusion Criteria:

* pregnancy
* patient's lack of consent to the examination

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
The utility of 18F-fluorocholine PET/CT in the imaging of parathyroid adenomas | 24 months
  Sensitivity and positive predictive value of 18F-FCH PET/CT in preoperative localisation of hyperfunctioning parathyroid tissue in patients with primary hyperparathyroidism

CONTACTS AND LOCATIONS:
Overall Officials: Andrzej Mazurek, MD, PhD, Principal Investigator — Military Institute of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cordellat IM. Hyperparathyroidism: primary or secondary disease? Reumatol Clin. 2012 Sep-Oct;8(5):287-91. doi: 10.1016/j.reuma.2011.06.001. Epub 2011 Oct 20. PMID 22089066
- [Result] Wilhelm SM, Wang TS, Ruan DT, Lee JA, Asa SL, Duh QY, Doherty GM, Herrera MF, Pasieka JL, Perrier ND, Silverberg SJ, Solorzano CC, Sturgeon C, Tublin ME, Udelsman R, Carty SE. The American Association of Endocrine Surgeons Guidelines for Definitive Management of Primary Hyperparathyroidism. JAMA Surg. 2016 Oct 1;151(10):959-968. doi: 10.1001/jamasurg.2016.2310. PMID 27532368
- [Result] Lopez-Mora DA, Sizova M, Estorch M, Flotats A, Camacho V, Fernandez A, Abouzian S, Fuentes-Ocampo F, Garcia JIP, Ballesteros AIC, Duch J, Domenech A, Duarte AM, Carrio I. Superior performance of 18F-fluorocholine digital PET/CT in the detection of parathyroid adenomas. Eur J Nucl Med Mol Imaging. 2020 Mar;47(3):572-578. doi: 10.1007/s00259-020-04680-7. Epub 2020 Jan 9. PMID 31919634